CLINICAL TRIAL: NCT03416647
Title: Superior Mesenteric Artery Syndrome: a Prospective Study in a Single Institution
Brief Title: SMAS: a Prospective Study in a Single Institution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, Angelica Ganss, Principal Investigator, Azienda Ospedaliera di Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOPadova
Record Dates: First submitted 2017-12-18; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Superior Mesenteric Artery Syndrome
Keywords: Superior Mesenteric Artery Syndrome; Chronic duodenal obstruction; Duodenojejunostomy; Wilkie's syndrome
MeSH Terms: conditions — Superior Mesenteric Artery Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMAS patients (Experimental)
  Interventions: Procedure: Duodenojejunostomy

INTERVENTIONS:
Procedure: Duodenojejunostomy — Duodenojejunostomy with or without duodenal resection

SUMMARY:
Superior Mesenteric Artery Syndrome (SMAS) is a rare cause of duodenal obstruction, that should be suspected in cases of chronic, refractory upper digestive symptoms. Between 2008 and 2016, 39 consecutive patients with chronic gastrointestinal symptoms and a diagnosis of SMAS were prospectively included in the study, in order to describe their demographic, clinical and outcome features. All patients underwent duodenojejunostomy.

ELIGIBILITY:
Inclusion Criteria (at least 2 of the following):

* severe and frequent upper digestive symptoms (occurring at least once a week), associated to poor quality of life and refractory response to medical treatment;
* a condition of underweight (BMI <18.5 kg/m2) associated with difficulty eating;
* severe complications of SMAS (e.g. gastric perforation, acute pancreatitis, aspiration pneumonia);
* suggestive findings of SMAS at barium swallow;
* diagnostic aortomesenteric angle and distance at CT/MR angiography.

Exclusion Criteria:

* inability to provide the informed consent;
* malignancies;
* bowel motility disorders;
* severe psychiatric illness;
* pregnancy;
* impossibility to perform the required diagnostic workup.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-10; Primary Completion 2016-05 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Symptom score | 47 months (IQR 34-72)
  Severity (0-6) + frequency (0-5) x 5 symptoms (abd pain, nausea, vomiting, reflux, bloating)
BMI | 47 months (IQR 34-72)
  Body mass index
Need for medical treatment | 47 months (IQR 34-72)
  PPIs, prokinetic drugs

CONTACTS AND LOCATIONS:
Overall Officials: Angelica Ganss, M.D., Principal Investigator — General Surgery Unit
Locations (1):
- General Surgery Unit, Padua, PD, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ganss A, Rampado S, Savarino E, Bardini R. Superior Mesenteric Artery Syndrome: a Prospective Study in a Single Institution. J Gastrointest Surg. 2019 May;23(5):997-1005. doi: 10.1007/s11605-018-3984-6. Epub 2018 Oct 5. PMID 30291587